CLINICAL TRIAL: NCT01334177
Title: Phase I Clinical Trial of VTX-2337, a Small Molecule Toll-Like Receptor 8 (TLR8) Agonist in Combination With Cetuximab in Patients With Recurrent or Metastatic Squamous Cell Carcinomas of the Head and Neck (SCCHN)
Brief Title: TLR8 Agonist VTX-2337 and Cetuximab in Treating Patients With Locally Advanced, Recurrent, or Metastatic Squamous Cell Cancer of Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7406; NCI-2011-00240 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 7406 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2011-03-21; First posted 2011-04-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — VTX-2337; Cetuximab; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (immunotherapy and monoclonal antibody therapy) (Experimental): Patients receive cetuximab IV over 60-120 minutes on days -28, -21, -14, -7 of weeks -4 to -1. Patients then receive cetuximab IV on days 1, 8, 15, and 22 and TLR8 agonist VTX-2337 SC on days 1, 8, 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: TLR8 agonist VTX-2337; Biological: cetuximab; Other: laboratory biomarker analysis; Other: pharmacogenomic studies

INTERVENTIONS:
Drug: TLR8 agonist VTX-2337 — Given SC
  Other Names: Toll-like receptor 8 agonist VTX-2337; VTX-2337
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study

SUMMARY:
This phase I trial studies the side effects and best dose of TLR8 Agonist VTX-2337 when given together with cetuximab in treating patients with locally advanced, recurrent, or metastatic squamous cell cancer of the head and neck (SCCHN). Biological therapies, such as TLR8 Agonist VTX-2337 may stimulate the immune system in different ways and stop tumor cells from growing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving TLR8 Agonist VTX-2337 together with cetuximab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability and to assess the dose-limiting toxicities (DLT) of VTX-2337 (TLR8 Agonist VTX-2337) when given in conjunction with cetuximab in order to define the maximum tolerated dose (MTD)/recommended phase II dose (RP2D).

SECONDARY OBJECTIVES:

I. To determine the pharmacodynamic immune response to VTX-2337 in combination with cetuximab.

II. Correlative assessments of immunologic response and activity will be performed, including: Quantitative evaluation of baseline immune status via in-vitro assessment of cytokine and chemokine response to immunostimulatory agents; quantitative assessment of plasma cytokines, chemokines, and other inflammatory markers via protein array; quantitative assessment of natural killer (NK) cells via flow cytometry; quantitative assessment of antigen-specific responses in cytokine-producing cells to common prognostic SCCHN antigens via interferon (INF)gamma-enzyme-linked immunosorbent spot (ELISpot).

III. To assess whether subjects with functional genetic variations in the TLR8 and FC-gamma-R IIIA genes have altered biological and/or clinical responses to VTX-2337, genetic characterization of subjects will be performed via standard genotyping assays.

TERTIARY OBJECTIVES:

I. To assess preliminary evidence of anti-tumor activity for the combination of VTX-2337 and cetuximab, as measured by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

OUTLINE: This is a dose-escalation study of TLR8 Agonist VTX-2337.

Patients receive cetuximab intravenously (IV) over 60-120 minutes on days -28, -21, -14, -7 of weeks -4 to -1. Patients then receive cetuximab IV on days 1, 8, 15, and 22 and TLR8 agonist VTX-2337 subcutaneously (SC) on days 1, 8, 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological or cytopathological confirmed diagnosis of squamous cell carcinoma of the head and neck region that is:

  * Locally advanced/recurrent and no longer amenable to local surgical or radiation therapy and/or
  * Has evidence of metastatic disease
* Patients may have been previously treated with systemic therapy but are otherwise deemed currently platinum-refractory, or would be deemed inappropriate or intolerant to platinum-based chemotherapy
* Patients must have completed definitive chemotherapy and/or radiation therapy >= 3 months prior to study entry
* Prior therapy with agents targeting/blocking the epidermal growth factor receptor (e.g. cetuximab and erlotinib) is allowable
* Performance Status: Eastern Cooperative Oncology Group (ECOG) 0 - 2
* Expected life expectancy of at least 12 weeks, as assessed by the Investigator
* Ability and willingness to comply with the study's visit and assessment schedule and to provide voluntary written informed consent
* Absolute neutrophil count (ANC) >= 1,500 cells/μL
* Platelet count >= 75,000 cells/μL
* Hemoglobin >= 8.0 g/dL
* Creatinine =< 2.0 mg/dL
* Total bilirubin =< 2.0 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]), serum glutamic pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN

  * For patients with liver metastases, AST, ALT < 5x ULN is acceptable
* Willingness to use a medically acceptable method of contraception throughout the study period and for 4 weeks after the final administration of VTX-2337 (all subjects)
* For female subjects with reproductive potential: a negative serum pregnancy test

Exclusion Criteria:

* Investigational therapy within 4 weeks of study entry
* Chemotherapy therapy or palliative radiation therapy within the previous 2 weeks prior to dosing with cetuximab or VTX-2337; patients should have recovered from major toxicities of prior therapy (If deemed reversible, toxicities should return to baseline or =< grade 2 in severity)
* Major surgery within the past 4 weeks prior to dosing with cetuximab or VTX-2337
* Concurrent symptomatic central nervous system (CNS) involvement, brain or leptomeningeal metastases; treated CNS involvement which has been stable > 28 days off systemic steroids may be included
* Major active psychiatric disorders which would limit compliance
* Treatment with oral or parenteral corticosteroids within 2 weeks prior to dosing with VTX-2337 or a requirement for systemic immunosuppressive therapy for any reason
* Active autoimmune disease
* Clinically significant cardiac disease (e.g., congestive heart failure, unstable or uncontrolled angina, myocardial infarction) within 6 months of dosing with VTX-2337
* Clinically significant ophthalmologic disease, defined as:

  * Current retinal vascular disorder, including active untreated diabetic retinopathy and/or
  * Previous or current uveitis
* Infection requiring parenteral antibiotic therapy or causing fever (temp > 100.5 degrees Fahrenheit [F] or 38.1 degrees Celsius [C]) within 1 week prior to dosing with VTX-2337
* Pregnant or breast-feeding females
* Uncontrolled inter-current illness, pre-planned surgery or procedure requiring hospitalization during the study period, or any other condition or circumstance that could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives
* Second primary malignancy that is clinically detectable (not including in situ carcinoma of the cervix, non-melanoma skin cancer or low-grade [Gleason score =< 6] localized prostate cancer) and demonstrating active progression at the time of consideration for study enrollment
* Known prior severe allergic/hypersensitivity to cetuximab or any of the components of the study treatment
* Known prior severe (>= Grade 3) rash and / or diarrhea toxicities to cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and the toxicities of TLR8 agonist VTX-2337 in combination with cetuximab | 28 days
  Frequency and severity of hematologic and non-hematologic adverse events will be compiled for each dose cohort. Assessment of adverse events will include type, incidence, severity (graded by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0), duration, seriousness, and relatedness; and clinically significant laboratory abnormalities.

SECONDARY OUTCOMES:
Pharmacodynamic immune response to TLR8 agonist VTX-2337 in combination with cetuximab | Day 1 of Course 1
  Will be predominantly descriptive with graphical information where available.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chow, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Dietsch GN, Lu H, Yang Y, Morishima C, Chow LQ, Disis ML, Hershberg RM. Coordinated Activation of Toll-Like Receptor8 (TLR8) and NLRP3 by the TLR8 Agonist, VTX-2337, Ignites Tumoricidal Natural Killer Cell Activity. PLoS One. 2016 Feb 29;11(2):e0148764. doi: 10.1371/journal.pone.0148764. eCollection 2016. PMID 26928328